CLINICAL TRIAL: NCT06196437
Title: Efficacy of Acupuncture on Catheter-Related-Bladder Discomfort After Transurethral Surgery： A Random Control Clinical Trial
Brief Title: Acupuncture for Catheter-Related-Bladder Discomfort After Transurethral Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Ran Pang, Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-109
Record Dates: First submitted 2023-12-07; First posted 2024-01-09 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Catheter-related-bladder Discomfort
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive acupuncture, five times per day form pre-operation to 3 days after operation. The selected acupoints include RN3,RN4, bilateral ST36,SP6,SP9 and LR3. All acupoints areas have been sterilized before acupuncture. needles (Ф0.30×50mm) will be directly inserted at a depth of 25-30 mm deep. Arrival of Qi by acupuncture and needle retaining for 20 minutes.
  Interventions: Other: Acupuncture
- Sham acupuncture (Sham Comparator): Participants will receive shame acupuncture, five times per day form pre-operation to 3 days after operation. The selected non-acupoints nearby RN3,RN4, bilateral ST36, SP6,SP9 and LR3, All acupoints areas have been sterilized before acupuncture. needles (Ф0.30×50mm) will be directly inserted at a depth of 5 mm deep. Needle retaining for 20 minutes and without needle manipulation.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Acupuncture — Participants will receive acupuncture.
  Arms: Acupuncture
Other: Sham Acupuncture — Participants will receive sham acupuncture.
  Arms: Sham acupuncture

SUMMARY:
The purpose of this study is to assess the effectiveness of acupuncture for treating catheter-related-bladder discomfort in adults after bladder outlet obstruction surgery.

DETAILED DESCRIPTION:
This randomized, controlled trial is aimed to assess the effectiveness of acupuncture in the treatment of catheter-related-bladder discomfort (CRBD) in adults after bladder outlet obstruction surgery. Eligible participants will be randomly allocated to acupuncture or sham acupuncture.

To minimize the evaluation bias, the outcome assessors and statisticians will be masked to treatment allocation besides participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old, signed informed consent
* Clinical diagnosis of bladder neck obstruction or benign prostatic obstruction
* Transurethral holmium laser resection of the prostate/transurethral cystoscopy posterior urethral decompression of the bladder neck was planned

Exclusion Criteria:

* Patients undergoing lower urinary tract surgery due to other diseases
* Complicated with urinary tract infection, urinary calculi, urethral stricture, neurogenic bladder, chronic interstitial cystitis
* Receiving treatment for other medical conditions that may affect bladder function
* Patients with severe heart, lung, cerebrovascular, liver, kidney, hematopoietic system and mental diseases
* Patients with contraindications to acupuncture treatment or fear acupuncture treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of CRBD | 24, 48, and 72 hours after surgery
  participants will wear an electronic counter to record the number of episodes of Catheter-Related-Bladder Discomfort (CRBD)
Severity of CRBD | 24, 48, and 72 hours after surgery
  participants will be requested to describe the situations of CRBD, the severity will be evaluated by the principal investigator. the scoring system for catheter- related bladder discomfort measurement as 4 levels: 0 score, no discomfort; 1 score, mild discomfort only reported upon questioning; 2 score, moderate discomfort, urge to pass urine reported by the patient without questioning; 3 score, severe discomfort, ruge to pass uine accompanied by behavioral responses, such as flailing limbs, storng verbal responses, or attempt to pull out the catheter. The higher scores means worse outcome.

SECONDARY OUTCOMES:
Incidence of moderate to severe CRBD | 24, 48, and 72 hours after surgery
  participants will wear an electronic counter to record the number of episodes of CRBD, they will be requested to describe the situations of CRBD, the severity will be evaluated by the principal investigator. The scoring system for catheter- related bladder discomfort measurement as 4 levels: 0 score, no discomfort; 1 score, mild discomfort only reported upon questioning; 2 score, moderate discomfort, urge to pass urine reported by the patient without questioning; 3 score, severe discomfort, ruge to pass uine accompanied by behavioral responses, such as flailing limbs, storng verbal responses, or attempt to pull out the catheter. The higher scores means worse outcome, 2 to 3 score would be identifited moderate to severe CRBD.
Lower urinary tract symptoms-IPSS | Before surgery, 1 week after surgery, and 12 weeks after surgery
  assessed by the International Prostate Symptom Score,(from 0 to 35score), the questionnaire includes 7 questions, the higher scores means worse outcome.
Lower urinary tract symptoms-OABSS | Before surgery, 1 week after surgery, and 12 weeks after surgery
  assessed by the Overactive Bladder Symptom Score,(from 0 to 15score), the questionnaire includes 4 questions, the higher scores means worse outcome.
Duration of indwelling catheter | At the time of catheter removal (assessed up to 7 days)
  by reviewing the clinical chart
Length of hospital stay | At the time of patient discharge (assessed up to day 14)
  by reviewing the clinical chart
Types of additional adjuvant drugs for CRBD | From date of randomization until the date of catheter removal , assessed up to 7 days
  by reviewing the clinical chart
Doses of additional adjuvant drugs for CRBD | From date of randomization until the date of catheter removal , assessed up to 7 days
  by reviewing the clinical chart
Postoperative quality of life was evaluated-PPBC | 24, 48, and 72 hours after surgery
  assessed by the Patient Perception of Bladder Condition (from 0 to 6score), the questionnaire includes 1 question, the higher scores means worse outcome.
Postoperative quality of life was evaluated- VAS | 24, 48, and 72 hours after surgery
  assessed by the visual analogue scale(from 0 to 10score), the questionnaire includes 1 question, the higher scores means worse outcome.
Postoperative quality of life was evaluated-QoL | 24, 48, and 72 hours after surgery
  assessed by the IPSS-quality of life(from 0 to 6score), the questionnaire includes 1 question, the higher scores means worse outcome.
uroflowmetry | Before surgery, 1 week after surgery, and 12 weeks after surgery
  uroflowmetry test

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China